CLINICAL TRIAL: NCT00495118
Title: Risperidone Depot (Microspheres) in the Treatment of Subjects With Schizophrenia or Schizoaffective Disorder - an Open-label Follow-up Trial of RIS-INT-62 and RIS-INT-85.
Brief Title: A Long-term Safety Study for Long-acting Injectable Risperidone in Schizophrenia or Schizoaffective Disorder Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002017
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; risperidone; intramuscular injection; long-acting injectable
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to document the long-term safety of 25, 37.5, or 50 mg long-acting injectable risperidone given via injection to the gluteal muscle every 2 weeks to subjects with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Noncompliance in taking medication is very common among people with schizophrenia, and is a frequent cause of relapse of symptoms. A long-acting injectable formulation that ensures slow but steady release of risperidone over a period of several weeks would eliminate the need to take medication on a daily basis, and improve compliance. This is an open-label, international, multicenter study in subjects with schizophrenia or schizoaffective disorder who completed the risperidone microspheres arm of study RIS-INT-62, or who completed study RIS-INT-85, or who dropped out of the risperidone microspheres arm of study RIS-INT-62 due to treatment with 75 mg long-acting injectable risperidone. Patients have to begin this study within 7 days of the final visit in the RIS-INT-62 or RIS-INT-85 studies. The end point visit of the RIS-INT-62 or RIS-INT-85 study serves as the first visit of this open-label study. Patients can start this study on the same dose as the last risperidone microsphere injection that they received in the previous study, or at a dose that was 12.5 mg lower or higher than the previously received dose. Patients who received 75 mg risperidone microsphere injection during study RIS-INT-62 can continue on this dose but an attempt will be made to decrease the dose to 50 mg within 3 months. The total study duration is planned to be at least 1 year or until approval of long-acting injectable risperidone in the respective country. The study hypothesis is that treatment with the long-acting injectable formulation of risperidone every 2 weeks for at least 1 year will be safe and well tolerated, as assessed by adverse event reporting, the extrapyramidal symptom rating scale, laboratory tests, vital signs measurements, physical examinations, body weight measurements, electrocardiograms, and injection site evaluations. Patients will receive injections of risperidone depot microspheres (25, 37.5, 50, or 75 mg) in their gluteal muscle at 2-weekly intervals for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (patients from RIS-INT-62 or RIS-INT-85) or schizoaffective disorder (patients from RIS-INT-62 only) according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria
* patient completed the risperidone microspheres arm of RIS-INT-62, or completed RIS-INT-85, or dropped out of the risperidone microspheres arm of RIS-INT-62 due to treatment with 75 mg long-acting injectable risperidone
* informed consent signed by the patient
* patient is otherwise healthy on the basis of a prestudy physical examination and medical history.

Exclusion Criteria:

* A DSM-IV Axis I diagnosis other than schizophrenia or schizoaffective disorder
* no pregnant or breast-feeding women
* no female patient of childbearing potential without adequate contraception
* no history of severe drug allergy or hypersensitivity
* no subjects known to be unresponsive to risperidone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2001-10; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To document the long-term safety of 25, 37.5 and 50 mg long-acting injectable risperidone from baseline until study end point.

SECONDARY OUTCOMES:
To document long-term efficacy by measuring mean values and clinical improvement in Positive and Negative Symptoms Scale (Visits 3 & 5 to 10), and Clinical Global Impression scale (Visits 2 to 10), compared with previous and extension baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- See also: A long-term safety study for long-acting injectable risperidone in schizophrenia or schizoaffective disorder patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=343&filename=CR002017_CSR.pdf